CLINICAL TRIAL: NCT04172922
Title: Treatment Protocol for the Use of the Topical Rapamycin/Sirolimus for Complicated Vascular Anomalies and Other Susceptible Lesions
Brief Title: Topical Rapamycin/Sirolimus for Complicated Vascular Anomalies and Other Susceptible Lesions
Acronym: NOVA
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: IRB suspended and subsequent early termination
Sponsor: Nemours Children's Clinic (Other)
Responsible Party: Principal Investigator, Craig Johnson, Radiology Chair, Nemours Children's Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NOVA0118
Record Dates: First submitted 2019-11-08; First posted 2019-11-21 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Vascular Anomaly
MeSH Terms: conditions — Vascular Malformations | interventions — Sirolimus

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Open label, topical sirolimus arm (Experimental): Single arm, open label study of1% sirolimus ointment applied to affected area twice daily for the first four weeks followed by once daily for 5 months.
  Interventions: Drug: Topical Sirolimus

INTERVENTIONS:
Drug: Topical Sirolimus — Open label, topical sirolimus (1%) cream will be applied to cutaneous component of complicated vascular anomalies twice daily for 4 weeks and once daily thereafter- for the duration of study.
  Other Names: rapamycin

SUMMARY:
Proposed Study: Treatment protocol for the use of the topical Rapamycin/Sirolimus for Complicated Vascular Anomalies and other susceptible lesions

1. Aim The aim of this treatment study is to evaluate the benefit and tolerability of topical sirolimus applied to cutaneous vascular anomalies in pediatric patients. The primary end point will be individually determined based on improvement in lesional clinical characteristics over baseline
2. Rationale for topical sirolimus use in VA The rationale for the use of topical sirolimus is to minimize these potential side effects and risks. Data for the use of topical sirolimus for vascular anomalies at this time are anecdotal and case reports only. As such, this prospective protocol seeks to determine the effectiveness and tolerability of topical sirolimus on patients with vascular anomalies that have a cutaneous component.
3. Experimental design This is an open-labeled efficacy trial with the aim to determine if topical sirolimus can be safe and efficacious in treating the cutaneous component of complicated vascular anomalies. Patients who meet eligibility criteria with a diagnosis of vascular anomaly (VA) with cutaneous component will be offered treatment with the investigational topical sirolimus. Patients will receive topical sirolimus therapy for a total of six months and will be monitored regularly at the research site for clinical response. Response will be based on pre-determined clinical criteria. Patients will be removed from study if there is no response at three months after initiation of therapy.

   Clinical response will be defined as improvement in measurable parameters defined at the time of initiation of therapy. These include
   1. Size of lesions, measured in two parallel longest diameters
   2. Flattening of lesion
   3. Number of vesicles
   4. Episodes of superinfection or bleeding
   5. Improvement in pain
4. Drug Information The topical sirolimus formulation will be made at a concentration of 1% sirolimus ointment. Bulk sirolimus powder will be compounded in a liposomal base in a GMP level pharmaceutical company. This base will enhance drug penetration into the skin. It ensures adequate adhesion to the application area and a low degree of systemic absorption. Due to limited absorption only mild side effects are expected.

DETAILED DESCRIPTION:
Patients with vascular anomalies (VA) have a spectrum of diseases that can be broadly classified into vascular tumors and malformations. Complicated vascular anomalies can cause disfigurement, chronic pain, and organ dysfunction with significant morbidity and mortality. Despite the severity of potential complications, we lack uniform guidelines for the treatment and response to treatment of children and young adults with these diseases. Pre-clinical and clinical data supporting the essential regulatory function of the PI3K/Akt/mTOR pathway in vascular growth and organization, and suggest a therapeutic target for patients with complicated vascular anomalies. Nemours Children's Hospital (NCH) and other groups have been successfully using the mTOR inhibitor siroli-mus in a selected group of patients with VA. NCH exclusively uses the systemic oral formulation of sirolimus. The potential toxicities of systemic sirolimus is well documented, and many patients do not tolerate systemic sirolimus. We hypothesize this study will advance our treatment options of vascular anomalies by offering topical sirolimus. This prospective open labeled study will allow us to determine the efficacy and tolerability of topical sirolimus in the treatment of complicated vascular anomalies. This will potentially generate data for the use of topical sirolimus as an alternative to systemic sirolimus for patients with complicated VA with a cutaneous component.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be more than 36 months and less than 21 years of age.
* Newly diagnosed with vascular anomalies (VA) or have a VA that failed therapy with systemic sirolimus or other systemic or surgical therapies.
* Patients who have undergone surgical resection or interventional radiology procedures for disease control are eligible to start topical sirolimus
* At least 2 weeks since undergoing any major surgery.
* Must not have received Myelosuppressive chemotherapy within 4 weeks of starting sirolimus.
* At least 7 days since the completion of therapy with a GF that supports platelet, red or white cell number or function.
* At least 14 days since the completion of therapy with a biologic agent.
* Patients with Kaposiform Hemagioendothelioma who have failed or are intolerant of systemic sirolimus therapy.
* Patients must not have received any non-FDA approved drug within 4 weeks or 5 half-lives, whichever is longer, prior to starting sirolimus and during treatment with sirolimus.
* XRT: > or = 6 months from involved field radiation to vascular tumor.
* Patients may not be currently receiving strong inhibitors of CYP3A4 and may not have received medications within 1 week of starting sirolimus.
* Patients may not be taking enzyme-inducing anticonvulsants, and may not have received these medications within 1 week of starting topical sirolimus, as these patients may experience different drug disposition.
* Adequate organ function
* Total bilirubin ≤1.5 x ULN for age
* SGPT (ALT) <5 x ULN for age
* Serum albumin > or = 2 g/dL.
* Fasting LDL cholesterol of <160 mg/dL
* Adequate Bone Marrow Function
* Hemoglobin > or = 8.0 gm/dL (may receive RBC transfusions)
* Platelet count > or = 50,000/microL (transfusion independent defined as not receiving a platelet transfusion within a 7 day period prior to sirolimus use)
* Adequate Renal Function
* A serum creatinine based on age
* Urine protein to creatinine ratio (UPC) < 0.3 g/l
* Karnofsky > or = 50 (>/=16 years of age) and Lansky >/ = 50 for patients < 16 years of age

Exclusion Criteria:

* Concurrent severe and/or uncontrolled medical disease which could compromise compliance with safety monitoring requirements for sirolimus (e.g. uncontrolled diabetes, uncontrolled hypertension, severe infection, severe malnutrition, chronic liver or renal disease, active upper GI tract ulceration).
* Chronic treatment with systemic steroids or another immunosuppressive agent.
* Patients who require medications that inhibit/induce CYP3A4 enzyme activity to control concurrent medical conditions.
* Known history of HIV seropositivity or known immunodeficiency.
* Women who are pregnant or breast feeding.
* Males or females of reproductive potential should agree to use an effective contraceptive method during the period they are receiving topical sirolimus and for 3 months thereafter.
* Patients unwilling or unable to comply with the safety monitoring requirements for sirolimus.
* Patients who currently have an uncontrolled infection, defined as receiving intravenous antibiotics.
* Patients with hemangioma
* Patients with symptomatic complicated vascular anomalies with severe systemic symptoms that will need systemic therapy.

Ages: 36 Months to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2024-02-15 (Actual); Study Completion 2024-02-15 (Actual)

PRIMARY OUTCOMES:
Reduction in Pain or local irritation | 24 weeks
  Response will be evaluated by physical exam and documented at 24 weeks of therapy.
Cyst formation | 24 weeks
  Response will be evaluated by physical exam and documented at 24 weeks of therapy.
Decrease in discharge | 24 weeks
  Response will be evaluated by physical exam and documented at 24 weeks of therapy.
Decrease in cyst formation | 24 weeks
  Response will be evaluated by physical exam and documented at 24 weeks of therapy.

SECONDARY OUTCOMES:
Sirolimus level | 24 weeks
  Sirolimus level in ng/ml.
Bilirubin level | 24 weeks
  Total bilirubin in mg/dL
Neutrophil level | 24 weeks
  Neutrophil count in mm3
ALT level | 24 weeks
  ALT level in units/liter
Serum Albumin | 32 weeks
  Serum Albumin level in g/liter
Fasting LDL | 24 weeks
  Fasting LDL level in mg/dl
Hemoglobin level | 24 weeks
  Hemoglobin level in g/dl
Platelet count | 24 weeks
  Platelet count in microliter
Urine Protein/creatinine | 24 weeks
  Urine Protein/creatinine levels in mL/min

OTHER OUTCOMES:
Changes in vital signs | 24 weeks
  Pre and Post vital signs evaluations (Pulse)Pulse, Respiration and Blood Pressure.
Temperature | 24 weeks
  Temperature in C/F
Respirations | 24 weeks
  Pre and Post vital signs evaluation (Respirations)
Blood pressure | 24 weeks
  Pre and Post vital signs evaluations (Blood pressure)
Changes in Weight | 24 weeks
  Weight will be collected in Kilograms.
Changes in Height | 24 weeks
  Height will be collected in meters
Changes in daily topical ointment applications | 24 weeks
  Medication diary(QOL) for Sirolimus topical ointment application documentation

CONTACTS AND LOCATIONS:
Overall Officials: Craig Johnson, DO, Principal Investigator — Nemours
Locations (2):
- United States (2):
  - Nemours Children's Health, Jacksonville, Jacksonville, Florida
  - Nemours Children's Hospital, Florida, Orlando, Florida